CLINICAL TRIAL: NCT02327143
Title: An Absolute Bioavailability Study of LY2835219 in Healthy Subjects Using the Intravenous Tracer Method
Brief Title: A Study of LY2835219 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15533; I3Y-MC-JPBS (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 200 mg LY2835219 (Experimental): 200 mg LY2835219 administered orally on day 1.
  Interventions: Drug: LY2835219
- 0.4 mg ¹³C₈-LY2835219 (Experimental): 0.4 mg ¹³C₈-LY2835219 given intravenously (IV) for 15 minutes, starting approximately 6 hours after the oral dose.
  Interventions: Drug: ¹³C₈-LY2835219

INTERVENTIONS:
Drug: LY2835219 — Administered orally
  Arms: 200 mg LY2835219
Drug: ¹³C₈-LY2835219 — Administered IV
  Arms: 0.4 mg ¹³C₈-LY2835219

SUMMARY:
The aim of this study is to compare how much of the study drug gets into the blood stream when it is given as a single oral dose and as an intravenous infusion (given directly into a vein via a small needle).

The study will also provide information on how well the study drug is tolerated when given as a capsule in combination with giving it intravenously, and information on any changes in heart function.

The study will last about 10 days. Screening is required within 28 days before study drug is given.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy sterile males or surgically sterile females or postmenopausal females
* Have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m^2)
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.
* Participants who are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have participated in a clinical trial involving investigational product within the last 90 days
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure
* Show evidence of human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have consumed any sensitive CYP2B6 substrate drugs, any CYP3A4 inhibitor or any CYP3A inducer, herbal supplements, grapefruits or grapefruit containing products, Seville oranges or Seville orange containing products, star fruits or star fruit containing products within 2 weeks prior to dosing or intend to consume during the study
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single arm study. Participants first received 200 mg LY2835219 and then 0.4 mg ¹³C₈-LY2835219 given 6 hours later.
Groups:
- 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219: 0.4 mg ¹³C₈-LY2835219 given intravenously (IV) for 15 minutes, starting approximately 6 hours after the oral dose on day 1.
Period: Day 1: Time 0 Hrs to 6 Hrs
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219
Started | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0
Period: Day 1: Time 6 Hrs - to Day 9
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219
Started | 0 | 11
Completed | 0 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- All Participants: 200 mg LY2835219 administered orally on day 1. 0.4 mg ¹³C₈-LY2835219 given intravenously (IV) for 15 minutes, starting approximately 6 hours after the oral dose on day 1.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.00 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Zero to Infinity [AUC(0-∞)] of LY2835219 and ¹³C₈-LY2835219
Time Frame: Predose, 2, 4, 6, 6.25, 6.5, 6.75, 7.25, 8.25,10, 12, 14, 24, 48, 72, 96,120, 144, 168,192 Hours Postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*h/milliliter (ng∙h/mL)
Groups:
- 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219: 0.4 mg ¹³C₈-LY2835219 given intravenously (IV) for 15 minutes, starting approximately 6 hours after the oral dose.
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219
Number analyzed (Participants) | 8 | 8
nanogram*h/milliliter (ng∙h/mL) | 3730 (31) | 15.4 (28)
Statistical Analysis 1: Comparison: 200 mg LY2835219 vs 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219; Test type: Superiority or Other; Ratio of geometric least squares = 0.448, 90% CI 2-sided [0.395 to 0.508] — Absolute bioavailability of LY2835219 following the administration of 200 mg LY2835219 (oral) with 0.4 mg [13C8]-LY2835219 (IV)

2. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of LY2835219
Time Frame: Predose, 2, 4, 6, 6.25, 6.5, 6.75, 7.25, 8.25,10, 12, 14, 24, 48, 72, 96,120, 144, 168,192 Hours Postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 200 mg LY2835219
Number analyzed (Participants) | 8
nanogram per milliliter (ng/mL) | 114 (32)

3. Secondary Outcome: PK: Time of Maximum Observed Drug Concentration (Tmax) of LY2835219
Time Frame: Predose, 2, 4, 6, 6.25, 6.5, 6.75, 7.25, 8.25,10, 12, 14, 24, 48, 72, 96,120, 144, 168,192 Hours Postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data
Measure: Median (Full Range); unit: hours
Arm/Group | 200 mg LY2835219
Number analyzed (Participants) | 8
hours | 6.63 [6.50 to 8.25]

ADVERSE EVENTS:
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg LY2835219 (N=11) | 200 mg LY2835219 + 0.4 mg ¹³C₈-LY2835219 (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days